CLINICAL TRIAL: NCT07226804
Title: Nanosecond Pulsed Field Ablation in the Management of Benign Thyroid Nodules
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0483; NCI-2025-08362 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Nodules; Pulsed Field Ablation
MeSH Terms: conditions — Thyroid Nodule | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — patient-reported outcomes questionnaire

SUMMARY:
To observe the outcomes of nsPFA therapy to treat benign thyroid nodules.

DETAILED DESCRIPTION:
Primary Objectives

• To evaluate the thyroid nodule volume changes over time in participants undergoing nsPFA as part of routine clinical care

Secondary Objectives

* To determine changes in health-related quality of life changes following ultrasound-guided nsPFA
* To evaluate the ultrasound features of thyroid nodules over time following ultrasound-guided nsPFA.
* To assess the incidence and nature of complications following ultrasound-guided nsPFA, categorized into Minor and Major complications.

ELIGIBILITY:
Eligibility Criteria

* Scheduled to undergo ultrasound guided nsPFA as standard of care
* Age 18 to 80 years.
* Capable of providing independent consent.
* Presence of biopsy-confirmed benign thyroid nodule , defined as one of the following:

  * Benign FNA X 2 or
  * Benign US guided FNA X 1 + benign thyroid nodule ultrasound appearance (TI-RADS 2) or
  * Benign FNA X 1 and radiographic/laboratory evidence of functional nature
* Nodule measuring >2cm in greatest dimension
* Presence of compressive symptoms reasonably attributable to thyroid nodule (i.e. pressure sensation, dysphagia, dysphonia, respiratory distress)
* No abnormal cervical lymph nodes during screening visit .

Exclusion Criteria

* Age <18
* Patients considered unsuitable for nsPFA by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04-26 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life Questionnaire | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Banuchi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org